CLINICAL TRIAL: NCT00930748
Title: Evaluation of the Potential of Endorectal MRI for the Staging and Recurrence of Prostate Cancer
Brief Title: Evaluation of MRI for Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: The MRI company forbidded additional scans with endorectal colil in this machine
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Orith Portnoy, Sheba Medical Center
Other Study IDs: SHEBA-08-4965-OP-CTIL
Record Dates: First submitted 2009-06-22; First posted 2009-06-30 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MR imaging with endorectal coil — MR imaging with endorectal coil
Device: MRI with endo-rectal coil — MRI with endo-rectal coil

SUMMARY:
The objective of this study is to evaluate imaging quality and correlation with histopathology in prostate cancer.

DETAILED DESCRIPTION:
The objective of this study is to evaluate of the potential of endorectal 3T MRI for the staging of prostate cancer before prostatectomy or recurrence of prostate cancer after prostatectomy

ELIGIBILITY:
Inclusion Criteria:

* Age of patients: up to 80 years.
* Men scheduled for radical prostatectomy due to prostate cancer or men post radical prostatectomy with suspicion of recurrence.
* Patients who are able and willing to give consent and able to have an MRI examination.

Exclusion Criteria:

* Contraindications to MRI including: claustrophobia, weight over 120 kg, implanted ferromagnetic materials or foreign objects, and known intolerance to the MRI contrast agent (e.g. Gadolinium or Dotarem)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during imaging (approximately 1 hr.)
* Any rectal pathology preventing probe insertion, (as active proctitis, active ulcerative colitis, fissure ani)
* Any spinal pathology that prohibits maintaining supine position for an hour
* Patients with documented myocardial infarction within one month of protocol entry, and patients with cardiac pacemakers
* Severe cerebrovascular disease (multiple CVA or CVA within 6 months)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
• MRI and pathology correlation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel